CLINICAL TRIAL: NCT02839096
Title: Once Daily Versus Twice Daily Iron Supplementation to Treat Anemia in Pregnancy: A Prospective, Randomized, Placebo Controlled, Double Blinded, Clinical Trial
Brief Title: Once Versus Twice Daily Iron Supplementation in Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds, PI left University
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Mistie Mills, Associate Professor, Ob/Gyn & Women's Health, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004638
Record Dates: First submitted 2016-06-09; First posted 2016-07-20 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Anemia in Pregnancy
MeSH Terms: interventions — Iron; ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Clinical Research Unit provides randomization order to the Investigational Pharmacy, which provides treatment or placebo tablets sets to the care provider.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Once Daily Dosing (Other): Randomized to 325mg of ferrous sulfate in the morning and placebo in the evening
  Interventions: Drug: Placebo; Drug: Ferrous Sulfate
- Twice Daily Dosing (Other): Randomized to 325mg of ferrous sulfate in the morning and 325mg of ferrous sulfate in the evening
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Placebo — Cellulose placebo that will be used in place of a second dose of ferrous sulfate in the subjects randomized to once daily dosing of ferrous sulfate
  Other Names: Iron
  Arms: Once Daily Dosing
Drug: Ferrous Sulfate — Subjects will receive once or twice daily dosing of ferrous sulfate. This will be provided by our hospital pharmacy and be identical in appearance to the placebo.
  Other Names: Iron

SUMMARY:
The investigators will randomize women diagnosed with anemia in the mid-trimester of pregnancy to once or twice daily iron supplementation

DETAILED DESCRIPTION:
Women defined as having iron deficiency anemia based on a low hemoglobin as defined by the American College of Obstetrics and Gynecology and a low serum ferritin, in the absence of hemoglobinopathy, will be randomized to ferrous sulfate 325mg PO daily or PO twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Iron deficiency anemia as defined by a Hgb of less than 11mg/dL in the first and 3rd trimester and 10.5mg/dL in the 2nd trimester and a serum ferritin of less than 15ug/mL.
* In accordance with American College of Obstetricians and Gynecologists (ACOG) guidelines, the Hgb cutoff will be reduced by 0.8mg/dL in African American women.
* In accordance with the standard of care, African American women and those with a mean corpuscular volume (MCV) on their routine screening complete blood count (CBC) of less than 70 will require a hemoglobin electrophoresis to exclude hemoglobinopathy prior to enrollment.

Exclusion Criteria:

* Multiple gestation
* Maternal hemoglobinopathy or hemochromatosis,
* Irritable bowel disease or irritable bowel syndrome
* History of bariatric surgery or extensive bowel surgery
* Individuals already receiving iron supplementation aside from prenatal vitamins.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mistie P Mills, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include (1) demographics, (2) baseline/postpartum hematocrit and levels of hemoglobin, ferritin and hepcidin, and (3) clinical data related to the pregnancy and outcomes. Protected personal information will be removed by trained staff at the Ob/Gyn Clinical Research Unit according to HIPAA guidelines. The final dataset will identify participants by a study number and dates will be replaced by time intervals. Data release is restricted to users under a data-transfer agreement (DTA) that provides for (1) a commitment to using the data only for research purposes and not to seek to identify any individual participant; (2) restrictions on redistribution of data to third parties, (3) a commitment to securing data using appropriate computer technology; and (4) a commitment to destroying or returning the data after analyses are completed. Upon DTA completion, access will be granted to a secured, cloud-based dataset monitored by the Information Technology Department.
Supporting Information: Study Protocol
Time Frame: Data will be available May 01, 2021 and will be available for 10 years from that date.
Access Criteria: 1. a commitment to using the data only for research purposes and not seek to identify any individual participant
  2. restrictions on redistribution of the data to third parties
  3. a commitment to securing the data using appropriate computer technology
  4. a commitment to destroying or returning the data after analyses are completed
  5. completion of a data-sharing agreement between the researcher requesting data and the University of Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Once Daily Dosing | Twice Daily Dosing
Started | 11 | 9
GI Questionnaire Data | 10 | 9
Delivery Data | 10 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Once Daily Dosing | Twice Daily Dosing | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.545 (3.959) | 29.333 (3.905) | 27.250 (4.290)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Baseline Hemoglobin [Mean (Standard Deviation); unit: g/dL] — Hemoglobin levels measured immediately prior to enrollment in the study. Population: One subject in the "Once Daily Dosing" delivered at a separate institution, so there is no delivery data for her.
  g/dL
    number analyzed (Participants) | 10 | 9 | 19
    (all) | 10.300 (0.645) | 11.000 (1.079) | 10.632 (0.924)
Baseline Hematocrit [Mean (Standard Deviation); unit: percent] — Hematocrit levels measured immediately prior to enrollment in the study. Population: One subject in the "Once Daily Dosing" delivered at a separate institution, so there is no delivery data for her.
  percent
    number analyzed (Participants) | 10 | 9 | 19
    (all) | 30.790 (1.608) | 32.480 (2.688) | 31.590 (2.292)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin
Description: Maternal Hemoglobin will be measured at baseline, at the time of admission for labor and delivery and on post partum day one. Postpartum day 1 hemoglobin was estimated from hematocrit by dividing by 2.941.
Time Frame: Change in hemoglobin from baseline to one day postpartum
Population: One participant delivered at another hospital and so baseline, but not delivery or postpartum hemoglobin measurements were obtained.
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Once Daily Dosing | Twice Daily Dosing
Number analyzed (Participants) | 11 | 9
g/dL
  change in hemoglobin from baseline to delivery: number analyzed (Participants) | 10 | 9
  change in hemoglobin from baseline to delivery | 0.51 [0.0176 to 1.002] | 0.656 [-0.054 to 1.365]
  baseline hemoglobin | 10.264 [9.895 to 10.632] | 11.000 [10.3622 to 11.638]
  hemoglobin at delivery: number analyzed (Participants) | 10 | 9
  hemoglobin at delivery | 10.810 [10.465 to 11.155] | 11.656 [11.077 to 12.235]
  estimated postpartum hemoglobin: number analyzed (Participants) | 10 | 9
  estimated postpartum hemoglobin | 10.105 [9.749 to 10.462] | 10.431 [9.629 to 11.233]
  change in hemoglobin from baseline to postpartum day 1: number analyzed (Participants) | 10 | 9
  change in hemoglobin from baseline to postpartum day 1 | -0.195 [-0.457 to 0.067] | -0.569 [-1.392 to 0.254]

2. Primary Outcome: Incidence of Gastrointestinal Side Effects (i.e. Constipation, Upset Stomach) as Measured by a Validated Questionnaire
Description: Record the incidence of gastrointestinal side effects (i.e. constipation, upset stomach) as measured by a validated questionnaire.
Time Frame: From enrollment to delivery, which will be an average of 10-12 weeks
Measure: Mean (95% Confidence Interval); unit: symptoms
Arm/Group | Once Daily Dosing | Twice Daily Dosing
Number analyzed (Participants) | 10 | 9
symptoms | 1.900 [0.828 to 2.972] | 1.222 [0.254 to 2.190]

3. Secondary Outcome: Incidence of Blood Transfusion at Delivery
Description: The number of patients who received a blood product transfusion at delivery.
Time Frame: At delivery
Measure: Number; unit: participants
Arm/Group | Once Daily Dosing | Twice Daily Dosing
Number analyzed (Participants) | 10 | 9
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Data were collected between enrollment and delivery, approximately 12 weeks.
Description: A questionnaire was administered to assess gastrointestinal symptoms. The incidence of one or more of nausea, hearburn, or abdominal pain is reported as a non-serious adverse event.
Arm/Group | Once Daily Dosing | Twice Daily Dosing
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 6/11 | 5/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Once Daily Dosing (N=11) | Twice Daily Dosing (N=9)
mild gastrointestinal symptoms (Gastrointestinal disorders) | 6 | 5 — A questionnaire used to assess GI symptoms included nausea, heartburn and abdominal pain. If any of these was reported a GI symptom was considered to have occurred

LIMITATIONS AND CAVEATS:
A sample size calculation predicted that 17 participants would be needed in each treatment arm. However, accrual was halted prematurely due to the move of the principal investigator to another institution. In total, 20 subjects were randomized in the study. The gastrointestinal symptom questionnaire was not completed by one subject and delivery data were not available for a separate subject, who did not deliver at the University of Missouri.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/96/NCT02839096/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT02839096/ICF_001.pdf